CLINICAL TRIAL: NCT02951949
Title: Exposure to Endogenous Estrogens and Imaging Parameters of Atherosclerosis Burden in Postmenopausal Women
Brief Title: Estrogen Exposure and Atherosclerosis in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Antonio Cano Sanchez, Full Professor Obstetrics and Gynecology, University of Valencia
Other Study IDs: Ayudas Fundación Eresa 2008
Record Dates: First submitted 2016-10-23; First posted 2016-11-01 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Atherosclerosis; Menopause; Estrogens; Carotid Intima-media Thickness; Coronary Stenoses; Women
Keywords: atherosclerosis, endogenous estrogens, age
MeSH Terms: conditions — Atherosclerosis; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Postmenopausal women: Postmenopausal women attending the outpatient service of a third level hospital for health control.

SUMMARY:
One hundred Spanish postmenopausal women accepted to be investigated for cardiovascular risk actors including clinical features, serum biochemical parameters, single nucleotide polymorphisms for estrogen receptor, and imaging parameters, carotid intima-media thickness (91 women) and coronary computed tomography (32 women). Multivariable analysis confirmed that both age and glucose level directly affected IMT. Estrogenic exposure, as measured by the allele associated with lower expression of the ER beta gene, was protective at the sinus and the wall. Findings at the coronary arteries, either moderate or high calcium index (CAC) and/or significant lumen stenosis were sporadic and did not allow for establishing association with any of the variables assessed.

DETAILED DESCRIPTION:
One hundred postmenopausal women living in the urban area of Valencia were invited to participate in a cross-sectional study in which a list of clinical and analytical risk factors for cardiovascular disease were assessed. Clinical factors included weight, waist circumference, body mass index and blood pressure. Analytical parameters included lipidogram, serum glucose and insulin, thyroid hormones (TSH and total T4), vitamin D, ultra-sensitive C-reactive protein, estradiol, and osteoprotegerin. Imaging studies were performed to identify the atherosclerotic burden at the carotid artery (intima-media thickness, measured by a high frequency ultrasound probe), and the coronaries (both coronary artery calcium(CAC) score and the degree of lumen stenosis). Genetic susceptibility was measured by studying single nucleotide polymorphisms of the estrogen receptor. The independent effect of each variable was analyzed with multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women free of previous diagnosis of cardiovascular disease, Caucasian ethnicity, urban origin, medium or medium-low socioeconomic extraction.

Exclusion Criteria:

* Previous diagnosis of cardiovascular disease, inability to understand the purpose and conditions of the study..

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women attending a clinical outpatient service in a third-level hospital for health control.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Carotid intima-media thickness. | 12 weeks
  Postmenopausal women attending clinical service for health control were measured carotid intima-media thickness by ultrasound.

SECONDARY OUTCOMES:
Changes in coronary calcium score. | 12 weeks
  Postmenopausal women attending clinical service for health control were measured the coronary calcium score with computed tomography.
Changes in coronary lumen stenosis. | 12 weeks
  Postmenopausal women attending clinical service for health control were measured the coronary lumen stenosis with computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cano, MD, Principal Investigator — University of Valencia
Locations (1):
- Hospital Clínico Universitario, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.